CLINICAL TRIAL: NCT06735378
Title: Exercise Preconditioning to Protect Against Dialysis-induced Cardiac Injury in Hemodialysis Patients: a Randomized Controlled Trial
Brief Title: Exercise Preconditioning to Protect Against Dialysis-induced Cardiac Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Nephrologist, Professor of Medicine, Medical Biophysics and Paediatrics, London Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 15393
Record Dates: First submitted 2024-11-26; First posted 2024-12-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hemodialysis; Cardioprotection
Keywords: Cardioprotection; Preconditioning Exercise; Hemodialysis

STUDY DESIGN:
Intervention Model Description: Open label, randomized, controlled, crossover trial with 2 conditions and 4 dialysis sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Randomization Order 1 (Experimental): Participants will be randomized into one of the two groups indicating the order in which they will receive the exercise intervention.
  Randomization Order 1 will receive the exercise treatment on the first day of the first week of the study. The other three days without exercise will consist of standard dialysis sessions with study procedures.
  Interventions: Other: Intradialytic Cycling
- Randomization Order 2 (Experimental): Participants will be randomized into one of the two groups indicating the order in which they will receive the exercise intervention.
  Randomization Order 2 will receive the exercise treatment on the first day of the fourth week of the study. The other three days without exercise will consist of standard dialysis sessions with study procedures.
  Interventions: Other: Intradialytic Cycling

INTERVENTIONS:
Other: Intradialytic Cycling — The impact of interdialytic exercise on cardio protection during HD has never been studied. This approach may enhance cardiovascular benefits and overall physical fitness, thereby contributing to better health outcomes in individuals undergoing HD.

SUMMARY:
The goal of this study is to determine what happens to the heart muscle contraction when people cycle before their hemodialysis treatment. Will pre-dialysis exercise protect the heart from a decrease in pumping of the heart muscle (called stunning) that can happen during hemodialysis. We will study whether pre-dialysis exercise decreases heart stunning, decreases the number and severity of symptoms commonly associated with hemodialysis, and other outcomes

DETAILED DESCRIPTION:
This will be the first randomized crossover-controlled trial with two experimental conditions assessing the impact of exercise preconditioning in the HD population. If proven effective exercise preconditioning could be developed as a therapeutic option to reduce rates of heart failure in the dialysis population.

ELIGIBILITY:
Inclusion Criteria:

* must be on chronic hemodialysis for at least 3 months
* age 18 years or older
* willing and able to provide informed consent
* assessed to be safe and able to exercise by unit HD Nephrologist

Exclusion Criteria:

* regular vigorous exercise outside of hemodialysis
* over 79 years of age
* intradialytic exercise < 3 months
* poor echogenicity
* acute coronary syndrome in the past 3 months
* unstable arrhythmia/angina
* shortness of breath at rest or with minimal activity
* symptomatic hypoglycemia (>2x/week in the week prior to enrolment)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of left ventricular segments undergoing a greater than 20% reduction in longitudinal strain as detected by echocardiogram | week 1 to week 4
  An echocardiogram will be completed pre-hemodialysis (HD) treatment and at peak hemodynamic stress (30 min before the end of HD treatment) at each of the four study sessions. Images will be captured in the left lateral position and standard apical 4, 2, and 3 chamber views will be recorded for analysis using automated speckle-tracking software (EchoPac, GE Healthcare)

SECONDARY OUTCOMES:
Evaluate potential targets of preconditioning by exercise-induced cardio protection by focusing on hemodynamics (Blood Pressure) | week 1 to week 4
  Systolic blood pressure (SBP), Diastolic blood pressure (DBP) and mean arterial pressure (MAP) will be measured using an automated blood pressure monitor integrated into the dialysis machine. Values will be monitored throughout each study.
Evaluate potential targets of preconditioning by exercise-induced cardio protection focusing on hemodynamics (CV Insight Monitoring), | week 1 to week 4
  The CV Insight contact device is a non-invasive continuous hemodynamic real time monitoring system used to assess cardiovascular and respiratory status using percutaneous photoplethysmography. The device will be attached to the right of the patient's forehead midline, approximately 2.5 cm above the level of the nose pre-dialysis and will remain intact until the patient is disconnected from the dialysis machine at each study session. Once attached, baseline recording will be obtained, and hemodynamic data will be continuously captured.
Evaluate potential targets of preconditioning by exercise-induced cardioprotection, focusing on hemodynamics (Finapres) | week 1 to week 4
  The Finometer utilizes a finger-cuff method to detect beat-to-beat changes in digital arterial diameter using an infrared photoplethysmography. The time-averaged data is subsequently downloaded to a computer-based analysis program for analysis. The finger-cuff will be placed on the participant's index finger at each study visit and will remain in place throughout the entire study visit
Evaluate potential targets of preconditioning by exercise-induced cardio protection, focusing on blood markers | week 1 to week 4
  Blood samples will be collected from the participants dialysis access. Before HD and at peak-stress of each study session, will be collected for biochemistry, proteomic analysis and translational approach.
Evaluate potential targets of preconditioning by exercise-induced cardio protection, focusing on erythrocyte deformability | week 1 to week 4
  Blood samples will be collected from the participants dialysis access. Before HD and at peak-stress of each study session for analysis of erythrocyte deformability which indicates microcirculation efficiency
Evaluate potential targets of preconditioning by exercise-induced cardio protection, focusing on endothelial function | week 1 to week 4
  Endothelial function is assessed by measuring the dilatory response of the brachial artery to increased blood flow generated by reactive hyperemia in the downstream forearm. At each study session participants are placed in the supine position and the brachial artery of the non-dominant arm, or the non-distended arm is scanned in longitudinal section using a 12 MHz linear transducer connected to a Vivid Q echograph (GE, USA) supplemented by an electrocardiogram (ECG).
Evaluate potential targets of preconditioning by exercise-induced cardioprotection, focusing on proteomic analysis. | week 1 to week 4
  Proteomic alterations in plasma are important in the inflammatory response to ischemia-reperfusion (IR) injury. Blood Samples (plasma) will be collected pre and peak dialysis at each study session for the analysis of changes induced by exercise preconditioning, with the aim of identifying new potential targets for cardio protection.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McIntyre, Principal Investigator — London Health Sciences Centre Research Institute
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Not yet determined
Supporting Information: Study Protocol
Time Frame: Not yet determined
Access Criteria: Not yet determined